CLINICAL TRIAL: NCT00927459
Title: A Placebo-Controlled, Single-Blind, Single-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of PRO-040201 in Male and Female Subjects With Hypercholesterolemia
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics (PK), and Pharmacodynamics (PD) of Liposomal siRNA in Subjects With High Cholesterol
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Potential for immune stimulation to interfere with further dose escalation.
Sponsor: Arbutus Biopharma Corporation (Industry)
Responsible Party: Mark Murray, PhD, CEO, Tekmira Pharmaceuticals Corporation
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TKM-ApoB-001
Record Dates: First submitted 2009-06-23; First posted 2009-06-25 (Estimated); Last update posted 2010-01-22 (Estimated); Status verified 2010-01

CONDITIONS: Hypercholesterolemia
Keywords: cholesterol; coronary artery disease
MeSH Terms: conditions — Hypercholesterolemia; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRO-040201 (Experimental): PRO-040201 with placebo control in each cohort
  Interventions: Drug: PRO-040201
- Placebo (Placebo Comparator): PRO-040201 with placebo control in each cohort
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRO-040201 — Single dose IV infusion
  Arms: PRO-040201
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
This study is a Phase 1, single-center, placebo-controlled, single-blind, first-in-human, single-ascending dose study in male and female subjects with high cholesterol. A maximum of 32 subjects is planned for enrollment in this study.

ELIGIBILITY:
Inclusion Criteria:

* Fasting, stable LDL-C ≥ 160 mg/dL
* Fasting, stable triglyceride < 400 mg/dL
* BMI between 22 and 35 kg/m2, inclusive
* Females must be of non-child bearing potential
* Males of reproductive potential must agree to practice effective contraception throughout the study and for 3 months following infusion

Exclusion Criteria:

* Clinically significant endocrine, hematologic, renal, hepatic, pulmonary, uncontrolled psychiatric, or neurologic disease
* Cancer within 5 years prior to screening
* History of congestive heart failure or chronic heart failure
* Uncontrolled cardiac arrhythmias
* History of coronary heart disease
* Clinically significant abnormal baseline ECG
* History of additional risk factors for torsades de pointes
* Hepatitis B, C, or HIV positive
* Current diagnosis or known history of liver disease
* A marked baseline prolongation of QT/QTc interval
* Known history of fibromyalgia, myopathy, myositis, rhabdomyolysis, any unexplained muscle pain, or a creatine phosphokinase (CPK) >3 x upper limit of normal (ULN) at screening
* Alanine aminotransferase, AST, GGT, or total bilirubin >2 x ULN at screening
* Serum creatinine > 1.5 mg/dL
* Systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg on 2 occasions during screening
* Concomitant use of medications that prolongs the QT/QTc interval
* Treatment with lipid lowering therapy within 30 days prior to screening
* Use of investigational drug within 3 months prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of PRO-040201 | 29 days

SECONDARY OUTCOMES:
Pharmacokinetics of PRO-040201 in Humans | 48 hours
Pharmacodynamics of PRO-040201 in Humans | 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Logan, MD, Principal Investigator — Medpace Clinical Pharmacology Unit
Locations (1):
- Medpace Clinical Pharmacology Unit, Cincinnati, Ohio, United States